CLINICAL TRIAL: NCT00610714
Title: A Phase II, Double-blind, Placebo-controlled, Multi-centre, Randomised Study of AZD0530 in Patients With Advanced Ovarian Cancer Sensitive to Platinum-based Chemotherapy
Brief Title: AZD0530 Phase II Study in Patients With Advanced Ovarian Cancer
Acronym: OVERT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8180C00015; AZD0530 Study 15
Record Dates: First submitted 2008-01-23; First posted 2008-02-08 (Estimated); Results first posted 2011-09-20 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Neoplasms; Ovarian Cancer
Keywords: Cancer; Tumour; Ovarian Neoplasms; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — saracatinib; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator (Active Comparator): carboplatin plus paclitaxel
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- 2 (Experimental): AZD0530 in combination with carboplatin plus paclitaxel
  Interventions: Drug: AZD0530; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: AZD0530 — oral once daily dose
  Arms: 2
Drug: Carboplatin — intravenous injection
  Other Names: CBDCA; Paraplatin®
Drug: Paclitaxel — intravenous infusion
  Other Names: Taxol®

SUMMARY:
The main purpose of this study is to determine if AZD0530 can improve the efficacy of standard chemotherapy for the treatment of ovarian cancer

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of advanced ovarian cancer
* Have evidence of recurrence or disease progression at least 6 months following treatment cessation of 1st or 2nd line platinum containing therapy
* Estimated life expectancy of more than 12 weeks

Exclusion Criteria:

* Central Nervous System (CNS) metastases
* Received more than 2 prior chemotherapy regimens for ovarian cancer treatment
* Inadequate bone marrow reserve
* Inadequate liver function, renal function or low haemoglobin
* Pregnant, breastfeeding or if of child-bearing status unwilling to use an acceptable method of contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Poole, Prof, Principal Investigator — Dept. of Oncology, University Hospital, Clifford Bridge Road, Walsgrave, Coventry; Mireille Cantarini, MD, Study Director — AstraZeneca
Locations (50):
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Herning
  - Research Site, Næstved
- France (10):
  - Research Site, Paris, Cedex 04
  - Research Site, Avignon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Pierre-Bénite
  - Research Site, Reims
  - Research Site, Vandœuvre-lès-Nancy
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, The Hague
- Norway (2):
  - Research Site, Bergen
  - Research Site, Oslo
- Research Site, Lima, Lima Province, Peru
- Portugal (4):
  - Research Site, Coimbra
  - Research Site, Funchal
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (4):
  - Research Site, Baia Mare, Maramureş
  - Research Site, Alba Iulia
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Russia (4):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Hospitalet Dellobregat(barcelo, Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Valencia, Valencia
- Research Site, Coventry, United Kingdom

REFERENCES:
- [Derived] Yap TA, Carden CP, Kaye SB. Beyond chemotherapy: targeted therapies in ovarian cancer. Nat Rev Cancer. 2009 Mar;9(3):167-81. doi: 10.1038/nrc2583. PMID 19238149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 58 cancer clinics in 12 countries (Bulgaria, Canada, Denmark, France, Netherlands, Norway, Peru, Portugal, Romania, Russia, Spain and UK) between April 2008 and March 2009.
Pre-assignment Details: Following enrolment there was a 28 day screening period, after which if all inclusion/exclusion criteria were met, patients were randomized to treatment.
Groups:
- AZD0530 , Paclitaxel , Carboplatin i.v.: AZD0530 175 mg in combination with Carboplatin AUC 6.0 mg/mL/min plus Paclitaxel 175 mg/m2 i.v.; Applies to the group receiving AZD0530 :An initial cohort of patients enrolled in the study were randomised to the 125 mg dose level; once confirmation of the tolerability of AZD0530 175 mg was available from a phase I dose escalation study (D8180C00023), all patients subsequently enrolled were randomised at the 175 mg dose level
- Carboplatin ,Paclitaxel: Carboplatin AUC 6.0 mg/mL/min, Paclitaxel 175 mg/m2 i.v;
Period: Overall Study
Arm/Group | AZD0530 , Paclitaxel , Carboplatin i.v. | Carboplatin ,Paclitaxel
Started | 105 | 106
Completed | 79 | 82
Not Completed | 26 | 24
Not completed — Adverse Event | 3 | 1
Not completed — Death | 12 | 18
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Study completion at 120 PFS events | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD0530 , Paclitaxel , Carboplatin i.v. | Carboplatin ,Paclitaxel | Total
Number analyzed (Participants) | 105 | 106 | 211
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (9.9) | 59.1 (10.2) | 58.265 (10.077)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 105 | 106 | 211
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 94 | 99 | 193
  Black | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Other | 8 | 4 | 12
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.758 (0.17) | 1.766 (0.206) | 1.762 (0.189)
World Health Organization (WHO) Performance Status [Number; unit: Participants] — minimum value=0=best outcome, maximum value=4=worst outcome
  Participants
    0 | 60 | 63 | 123
    1 | 41 | 42 | 83
    2 | 4 | 1 | 5
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
Primary Tumour Location (Number of Participants) [Number; unit: Participants]
  Ovary | 98 | 98 | 196
  Peritoneum | 4 | 5 | 9
  Uterine/fallopian tube | 3 | 1 | 4
  Site cannot be determined | 0 | 1 | 1
  Unavailable | 0 | 1 | 1
Tumour Grade [Number; unit: Participants]
  Well Differentiated (G1) | 8 | 8 | 16
  Mod. Differentiated (G2) | 29 | 25 | 54
  Unavailable (G3) | 45 | 53 | 98
  Undifferentiated (G4) | 4 | 6 | 10
  Unassessable (GX) | 15 | 14 | 29
  Missing | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Evaluated by Response Evaluation Criteria In Solid Tumors ( RECIST)
Description: Number of responders (complete (CR) or partial (PR) responders). CR = disappearance of all target lesions PR = 30% decrease in the sum of the longest diamete. Analysis was based on August 31, 2009 data cut-off , and was performed with patients who had measurable disease and received AZD0530 175mg or Placebo 175mg.
Time Frame: Response is evaluated from randomization to objective disease progression per RECIST criteria or death due to any cause in the absence of progression (conducted when a minimum of 78 progression free survival events had occurred)
Measure: Number; unit: Participants
Arm/Group | AZD0530 , Paclitaxel , Carboplatin i.v. | Carboplatin ,Paclitaxel
Number analyzed (Participants) | 88 | 87
Participants | 47 | 45

2. Secondary Outcome: Progression-free Survival (PFS) as Evaluated by RECIST
Description: Interval between date of randomization and earliest date of objective disease progression per RECIST criteria or death due to any cause in the absence of progression. Analysis was based on August 31, 2009 data cut-off (78 PFS events analysis) and was performed with patients in ITT analysis set who received AZD0530 175mg or Placebo 175mg.
Time Frame: Date of randomization to earliest date of objective disease progression or death due to any cause (conducted when a minimum of 78 progression free survival events had occurred)
Measure: Median (Full Range); unit: Months
Arm/Group | AZD0530 , Paclitaxel , Carboplatin i.v. | Carboplatin ,Paclitaxel
Number analyzed (Participants) | 96 | 93
Months | 8.28 [0 to 11.04] | 7.79 [0.72 to 12.12]

3. Secondary Outcome: Overall Survival (Number of Deaths)
Description: Interval between date of randomization and death due to any cause. Analysis was based on January 31, 2010 data cut-off and was performed with patients in ITT analysis set who received AZD0530 175mg or Placebo 175mg. At this time, data were still immature and median overall survival was not reached. Number of deaths is presented instead
Time Frame: Date of randomization to death due to any cause
Measure: Number; unit: Participants
Arm/Group | AZD0530 , Paclitaxel , Carboplatin i.v. | Carboplatin ,Paclitaxel
Number analyzed (Participants) | 96 | 93
Participants | 12 | 14

ADVERSE EVENTS:
Arm/Group | AZD0530 , Paclitaxel , Carboplatin i.v. | Carboplatin ,Paclitaxel
Serious Adverse Events (participants affected / at risk) | 46/105 | 26/106
Other Adverse Events (participants affected / at risk) | 102/105 | 104/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0530 , Paclitaxel , Carboplatin i.v. (N=105) | Carboplatin ,Paclitaxel (N=106)
Febrile Neutropenia (Blood and lymphatic system disorders) | 14 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal Fistula (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 1
Asthenia (General disorders) | 2 | 0
Drug Hypersensitivity (Immune system disorders) | 4 | 5
Anaphylactic Shock (Immune system disorders) | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Abdominal Wall Abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Device Related Sepsis (Infections and infestations) | 1 | 0
Enteritis Infectious (Infections and infestations) | 1 | 0
Escherichia Infection (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 1 | 0
Blood Creatinine Increased (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin Decreased (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hot Flush (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD0530 , Paclitaxel , Carboplatin i.v. (N=105) | Carboplatin ,Paclitaxel (N=106)
Neutropenia (Blood and lymphatic system disorders) | 45 | 38
Anaemia (Blood and lymphatic system disorders) | 40 | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 28 | 31
Leukopenia (Blood and lymphatic system disorders) | 17 | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 0
Nausea (Gastrointestinal disorders) | 68 | 64
Diarrhoea (Gastrointestinal disorders) | 44 | 36
Vomiting (Gastrointestinal disorders) | 43 | 39
Constipation (Gastrointestinal disorders) | 27 | 30
Abdominal Pain (Gastrointestinal disorders) | 15 | 22
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 10
Stomatitis (Gastrointestinal disorders) | 6 | 10
Fatigue (General disorders) | 37 | 42
Asthenia (General disorders) | 36 | 30
Pyrexia (General disorders) | 22 | 11
Oedema Peripheral (General disorders) | 3 | 9
Mucosal Inflammation (General disorders) | 6 | 7
Malaise (General disorders) | 3 | 6
Drug Hypersensitivity (Immune system disorders) | 16 | 24
Nasopharyngitis (Infections and infestations) | 8 | 15
Urinary Tract Infection (Infections and infestations) | 11 | 9
Cystitis (Infections and infestations) | 8 | 2
Weight Decreased (Infections and infestations) | 6 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 33 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 25
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 13
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 9
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 9
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Peripheral Sensory Neuropathy (Nervous system disorders) | 28 | 26
Neuropathy Peripheral (Nervous system disorders) | 17 | 24
Headache (Nervous system disorders) | 9 | 14
Paraesthesia (Nervous system disorders) | 8 | 14
Dizziness (Nervous system disorders) | 5 | 11
Dysgeusia (Nervous system disorders) | 8 | 6
Anxiety (Psychiatric disorders) | 1 | 15
Insomnia (Psychiatric disorders) | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 55 | 64
Rash (Skin and subcutaneous tissue disorders) | 15 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 9
Erythema (Skin and subcutaneous tissue disorders) | 7 | 3
Hypertension (Vascular disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites.